CLINICAL TRIAL: NCT00926666
Title: A Dose Finding Study for Ultrasound Guided Anterior Psoas Compartment Blocks in Patients With a Fractured Neck of Femur?
Brief Title: A Dose Finding Study for Pain Relief of a Broken Hip
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Dr aureen Travers / R+D Cooridator, NHS Greater Glasgow and Clyde
Allocation: Non-Randomized | Model: Single Group | Masking: Triple
Other Study IDs: MW001; EURACT 2009-013462-25; R+D:NumberGN09AN334
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Femoral Neck Fractures
Keywords: Ageing; Pain; Pharmacology; Imaging; Anaesthesiology; Musculoskeletal disease
MeSH Terms: conditions — Femoral Neck Fractures; Pain; Musculoskeletal Diseases | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Levobupivacaine — Dose finding study for levobupivacaine in fractured neck of femur patients. Ultrasound guided anterior psoas compartment nerve block to determine EC50 using up/Down methodology in patient before surgery to fix broken hip.

SUMMARY:
Studies have suggested a link with effective pain relief and reduced illness and death in high risk patients. Ultrasound guided nerve blocks have been associated with an increased success rate and allow visualization of all the anatomical structures and the distribution of the local anesthetic on injection. The hospital mortality for patients admitted to hospital from home in the UK in 2006 with a fractured hip is 14.3% (Bottle and Aylin 947-51).

The aim of this clinical trial is to determine the effective dose of local anesthetic to provide pain relief to patients with a broken hip using ultrasound to guide needle insertion. The hospital mortality for patients admitted to hospital from home in the UK in 2006 with a fractured hip was 14.3%. Patients for emergency surgical fixation or replacement of broken hip will be recruited prior to surgical fixation. All patients recruited to this study will receive standard anesthesia and surgical fixation of their broken hip.

The trial can be divided into two sequential parts; the results of part A will be an amount of local anesthetic which will relieve pain of a broken hip in 95% of all patients. Part B will determine the duration of pain relief provided by the amount of local anaesthetic from part A and blood levels of local anesthetic.

In parts A and B a standard pain relieving nerve block to numb the nerves supplying the hip joint will be administered using ultrasound to guide the injection of local anesthetic. The patient will then be observed for 30 minutes during which time the feeling in the upper leg and pain scores will be recorded. Patients with ineffective nerve blocks will be given immediate pain relief and withdrawn from further participation in the study.

In part A the amount of local anesthetic for the next patient will be increased or decreased if the nerve block is ineffective or effective respectively.

In part B the dose will be the same (calculated from the results of part A). In order to determine the duration of pain relief pain scores will be recorded hourly for up to 24 hours. Blood samples will be taken before the pain relieving nerve block and at 5, 10, 20, 30 and 60 minutes afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Emergency proximal fractured neck of femur for surgical fixation
* Visual analogue pain score at rest of >=5
* American Society of Anaesthesiology grading <=4
* Able to give informed consent
* Resting visual analogue pain score of greater than 50mm on a 100mm scale before recruitment
* Patient is able to cooperate with sensory testing of lower limb function

Exclusion Criteria:

* Abnormal clotting screen (coagulopathy) or thrombocytopenia (< 100,000)
* Acute mental test score of <=7 at any time preoperatively
* Allergy to local anaesthetic
* Contra-indication to levobupivacaine
* Signs, symptoms or laboratory evidence of local infection or systemic sepsis
* No pre-existing neurological deficit (sensory or motor) affecting the lower limb
* Patient with lower limb amputations or other condition affecting sensation in lower limbs
* Patient with a history of chronic pain

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours after local anaesthetic nerve block

SECONDARY OUTCOMES:
VAS resting acute pain scores | 10 mins, 20 mins and 30 mins after nerve block
Blood pressure, respiratory rate, pulse and oxygen saturations | 10 mins, 20 mins and 30 mins after nerve block
Liver function tests | Before nerve block
Venous blood gases | before nerve block
Serum levels of levobupivacaine | At 5, 10, 20, 30 and 60 mins after nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J Watson, MB chB, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Western Infirmary, Glasgow, Lanarkshire, United Kingdom